CLINICAL TRIAL: NCT03834753
Title: A Clinical Effectiveness, Multicenter, Randomized, Double-masked, Controlled Study of the Efficacy and Safety of ONS-5010 in Subjects With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration
Brief Title: A Clinical Effectiveness Study Examining the Efficacy and Safety of ONS-5010 in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Outlook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONS-5010-002
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration; Wet Macular Degeneration
Keywords: Subfoveal Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bevacizumab (Experimental): ONS-5010
  Interventions: Biological: bevacizumab
- ranibizumab (Active Comparator)
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: bevacizumab — 1.25 mg, intravitreal injection
  Other Names: ONS-5010
  Arms: bevacizumab
Biological: ranibizumab — 0.5mg, intravitreal injection
  Arms: ranibizumab

SUMMARY:
This research study will examine the safety and effectiveness of ONS-5010 in participants with AMD. The goal is to prevent vision loss by evaluating the effectiveness of ONS-5010 as compared with ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Active primary Subfoveal Choroidal Neovascularization lesions secondary to Age-related macular degeneration (AMD) in the study eye
* Best corrected visual acuity of 25-67 letters read (20/50 to 20/320 Snellen equivalent)
* Study eye must:

  * Have active leakage on Fluorescein Angiogram involving the fovea
  * Have edema involving the fovea
  * Be free of scarring, fibrosis, or atrophy involving the central foveal zone

Exclusion Criteria:

* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1-month preceding randomization
* Any concurrent intraocular condition in the study eye that may require medical or surgical intervention or contribute to vision loss within 1 year
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous haemorrhage in the study eye
* Polypoidal choroidal vasculopathy (PCV) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Current treatment for active systemic infection
* Known allergy to any component of the study drug or history of allergy to fluorescein , not amenable to treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who gain 15 or more letters in best corrected visual acuity (BCVA) | Baseline, 11 months
  BCVA to be assessed as letters read using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts. A positive change represents an improvement in visual acuity.

SECONDARY OUTCOMES:
Mean change in the best corrected visual acuity | Baseline, monthly to 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who gain at least 10 letters in the best corrected visual acuity | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who gain at least 5 letters in the best corrected visual acuity | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who lose fewer than 15 letters in the best corrected visual acuity | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A negative change represents a decrease in visual acuity.
Proportion of participants with visual-acuity Snellen equivalent of 20/200 or worse | Baseline, 11 months
Percentage of participants with ocular adverse events, non-ocular adverse events, grade 3 and above laboratory abnormalities, and vital sign abnormalities | 11 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Kissner, PhD, Study Director — Outlook Therapeutics, Inc.
Locations (49):
- United States (49):
  - Clinical Site, Tucson, Arizona
  - Clinical Site, Arcadia, California
  - Clinical Site, Beverly Hills, California
  - Clinical Site, Campbell, California
  - Clinical Site, Glendale, California
  - Clinical Site, Laguna Hills, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Mountain View, California
  - Clinical Site, Oxnard, California
  - Clinical Site, Palm Desert, California
  - Clinical Site, Poway, California
  - Clinical Site, Sacramento, California
  - Clinical Site, Santa Maria, California
  - Clinical Site, Tustin, California
  - Clinical Site, Golden, Colorado
  - Clinical Site, Hamden, Connecticut
  - Clinical Site, Clearwater, Florida
  - Clinical Site, Pinellas Park, Florida
  - Clinical Site, Sarasota, Florida
  - Clinical Site, Winter Haven, Florida
  - Clinical Site, Augusta, Georgia
  - Clinical Site, Marietta, Georgia
  - Clinical Site, Downers Grove, Illinois
  - Clinical Site, Lemont, Illinois
  - Clinical Site, Springfield, Illinois
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Hagerstown, Maryland
  - Clinical Site, Edina, Minnesota
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Bloomfield, New Jersey
  - Clinical Site, Albuquerque, New Mexico
  - Clinical Site, New York, New York
  - Clinical Site, Chambersburg, Pennsylvania
  - Clinical Site, Monroeville, Pennsylvania
  - Clinical Site, Rapid City, South Dakota
  - Clinical Site, Germantown, Tennessee
  - Clinical Site, Abilene, Texas
  - Clinical Site, Amarillo, Texas
  - Clinical Site, Arlington, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Grapevine, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, McAllen, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, The Woodlands, Texas
  - Clinical Site, Willow Park, Texas
  - Clinical Site, Salt Lake City, Utah
  - Clinical Site, Norfolk, Virginia
  - Clinical Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Data will not be shared until all global regulatory filings are complete.